CLINICAL TRIAL: NCT00803426
Title: Ultrasound Guided Popliteal Fossa Block. Does Blockade Distal to Sciatic Nerve Bifurcation Speed Onset Time? A Prospective, Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-0495-B
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2009-07

CONDITIONS: Ankle/Foot Surgery
Keywords: ultrasound-guided regional anesthesia; nerve block; popliteal fossa; sciatic nerve; common peroneal nerve; tibial nerve; onset time; ankle surgery; foot surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Local anesthetic will be injected above the division of the sciatic nerve.
  Interventions: Procedure: Sciatic nerve blockade for ankle/foot surgery
- 2 (Experimental): Local anesthetic will be injected below the division of the sciatic nerve, around the common peroneal and tibial nerves.
  Interventions: Procedure: Sciatic nerve blockade for ankle/foot surgery

INTERVENTIONS:
Procedure: Sciatic nerve blockade for ankle/foot surgery — Injection of local anesthetic near the nerve to achieve anesthesia.

SUMMARY:
Sciatic nerve block is used routinely in ankle and foot surgery. It is applied often by a posterior approach at the popliteal fossa, near where the nerve divides into the common peroneal and tibial nerves. Due to the size of the sciatic nerve, the largest in the body, infiltration of anesthetic and onset of anesthesia can take a significant amount of time. This study hypothesizes that selectively blocking both the common peroneal and the tibial nerves distal to the bifurcation may result in a faster block onset than blockade of the sciatic nerve proximal to its bifurcation.

DETAILED DESCRIPTION:
Sciatic nerve block (SNB) has been shown to reduce postoperative pain and opioid requirements, as well as improve patient satisfaction after outpatient foot and ankle surgery. The sciatic nerve divides into two terminal branches (the common peroneal and tibial nerves) in the popliteal fossa. Through these two branches it innervates the entire leg, ankle and foot except for the skin over the anterior-medial aspect of the leg, which is supplied by the saphenous nerve, a branch of the femoral nerve.

Many approaches have been described to sciatic nerve blockade. High in the thigh or buttock are the classical posterior approach, the supine approach, and the anterior approach. In the popliteal fossa, a posterior, a lateral and a medial approach have been described. The popliteal fossa approaches are most commonly used to provide regional anesthesia and/or analgesia for major foot and ankle surgery.

Traditional nerve localization techniques include seeking paresthesiae on needle to nerve contact, or alternatively seeking a muscle response to electrical nerve stimulation using a blunt insulated needle and a peripheral nerve stimulator. However, block results with traditional nerve localization techniques are highly variable, often requiring high local anesthetic doses, and a prolonged onset time. When a distal approach in the popliteal fossa is used (5-7 cm above the knee crease) with a nerve stimulator technique, a double motor response (both tibial and peroneal components) may be required to achieve consistent success.

Recently, ultrasound guided techniques for SNB at the popliteal fossa have been described. Ultrasound guidance offers the unique advantages of real time anatomic assessment of the sciatic nerve itself, its site of bifurcation, and its relationship to surrounding muscles and the popliteal vessels. In a recent study we have shown that ultrasound guidance significantly improves the success rate of SNB at the popliteal fossa via a posterior approach.

Despite these advantages, a prolonged onset time for complete blockade of up to 30-60 minutes (depending on the choice and dose of local anesthetic) is common. This may be a limitation to the widespread use of popliteal sciatic nerve blockade in a peri-operative environment, where a faster block onset may be preferable. This delayed onset has been attributed to the large size of the sciatic nerve. Therefore logically it should be faster to induce a block by depositing the local anesthetic after the sciatic nerve divides where the connective tissues decrease and the nerves are superficial. No exact mathematical data is available looking into onset times for nerves with varying diameter, as no previous studies are done in this area.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-III
2. 18-85 years of age, inclusive
3. 50-120 kg, inclusive
4. 150 cm of height or grater Scheduled for major elective foot or ankle surgery for which sciatic nerve block is indicated

Exclusion Criteria:

1. Contraindications to sciatic nerve block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the popliteal area)
2. Significant peripheral neuropathy or neurological disorder affecting the lower extremity
3. Pregnancy
4. History of alcohol or drug dependency/abuse
5. History of significant psychiatric conditions that may affect patient assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Onset time of anesthesia. | every 5 minutes until start of surgery

SECONDARY OUTCOMES:
Block procedure time, complications, location of the sciatic nerve bifurcation, postoperative pain, patient satisfaction with pain control | up to 2 days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada